# PARTICIPANT INFORMATION SHEET TEMPLATE FOR ADULTS



**Postoperative Pain After Caesarian Section** 

**NCT** number:

Date: 03 October 2022

# INVITATION TO PARTICIPATE IN A RESEARCH PROJECT

# WOULD YOU LIKE TO PARTICIPATE IN A RESEARCH PROJECT ABOUT PAIN, NAUSEA AND PRURITUS AFTER SPINAL ANAESTHESIA?

You are invited to participate in a research project where we will measure pain, nausea and pruritus after undergo caesarean section. You have been asked to participate in this study because you are a woman planning a caesarean section.

#### WHAT IS THE PROJECT ABOUT?

This is a request for you to participate in a study to examine pain, nausea and pruritus during the first 24 hours following the operation. We will also measure the amount of additional analgetics you receive, what type and medication against nausea. This is to evaluate if the current pain management at our hospital should be adjusted, for example adding morphine to the spinal anaesthesia.

You are invited because you will undergo caesarean section in spinal anaesthesia. We will examine how much pain and nausea you experience the first 24 hours. We will ask about pain and nausea according to a table. A nurse/midwife will record your answers every 30 minutes at the postoperative care unit, and every 4 hours at the maternity ward.

#### FORESEEABLE BENEFITS AND PREDICTABLE RISKS AND BURDENS OF TAKING PART

Advantages by participating in our project is that you will receive close follow up and we will know more about how you are doing after the caesarean section.

The disadvantage is that we will ask you about symptoms regularly.

### VOLUNTARY PARTICIPATION AND THE POSSIBILITY TO WITHDRAW CONSENT

Participation in the project is voluntary. If you wish to take part, you will need to sign the declaration of consent on the last page. You can, at any given time and without reason withdraw your consent. This will not have any consequences for any future treatment

If you choose not to participate, you will still receive the same treatment and the same level of observation.

If you decide to withdraw participation in the project, you can demand that your personal data concerning health be deleted, unless however, the personal data concerning health and tests have already been analysed or used in scientific publications. If you at a later point, wish to withdraw consent or have questions regarding the project, you can contact section chief physician Jorunn Korneliussen, contact information at the bottom.

#### WHAT WILL HAPPEN TO YOUR PERSONAL DATA CONCERNING HEALTH?

Any personal data concerning health that has been recorded about you will only be used as described in the purpose of the project. You have the right to access information that has been recorded about you and the right to stipulate that any error(s) in the information that is recorded is/are corrected. You also have the right to know which security measures have been/will be taken when your personal data concerning health is processed.

All information will be processed and used without your name or personal identification number, or any other information that is directly identifiable to you. A code links you and your personal data concerning health via an identifier list. Only project manager Conrad Bjørshol and section chief physician Jorunn Korneliussen will have access to the information.

Information about you will be anonymised and planned to be used by 31.12. 22. For control purpose we will keep the information on an approved research server until 32.12.2027, after that they will be deleted.

#### **INSURANCE**

Patient Injuries Act

#### **FINANCE**

Research group will receive payment form their employer. There are no sponsorship funds.

#### **APPROVAL**

The Regional Committee for Medical and Health Research Ethics has reviewed and approved the Research Project case number 194475

In accordance with the General Data Protection Regulation the controller Stavanger Universitetssykehus and the project manager Conrad Bjørshol is independently responsible to ensure that the processing of your personal data concerning health has a legal basis.

The processing of personal data is in accordance with REK (Regional ethical comitee) with case number 194475 and PVO (Data protection officer) at SUS ref. ID 1399.

You have the right to submit a complaint on the processing of your personal health data concerning health to the Norwegian Data Inspectorate (Datatilsynet).

## CONTACT INFORMATION

If you have any questions regarding the research project, you can get in touch with

Jorunn Korneliussen, Section chief physician.

Mail address: korj@sus.no Mobile phone: 90470706

# [Insert Project Title, Date and Version number here]

You can also get in touch with the Institution's Data Protection Officer (personvernombud) if you have any questions related to the use of your personal health data concerning health in the research project personvernombudet@sus.no.

# [Insert Project Title, Date and Version number here]

I CONSENT TO PARTICIPATING IN THE RESEARCH PROJECT AND THAT MY PERSONAL DATA CONCERING HEALTH AND BIOLOGICAL MATERIAL CAN BE USED AS DESCRIBED ABOVE

| [Remove the alternative(s) that are not applicable] | |
|---|---|
| City/Town and date | Participant's Signature |
| | Participant's Name (in BLOCK LETTERS) |
| I confirm that I have given informatio only in the instances where the inform | n about the research project [You can include this sentence if you wish, nation is given face to face.] |
| Place and date | Signature |
| | Role in the research project |